CLINICAL TRIAL: NCT04095338
Title: Assistive Robotic in the Elderly: Innovative Models in the Rehabilitation of the Elderly With Hip Fractures Through Technological Innovation
Brief Title: Innovative Models in the Rehabilitation of the Elderly With Hip Fractures Through Technological Innovation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INRCA_03_2019
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Hip Fractures; Frail Elderly; Robotic Rehabilitation
Keywords: hip fracture; rehabilitation; robotics
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Ten traditional physical treatment sessions divided into 2 training sessions per week for 5 weeks
  Interventions: Other: traditional rehabilitation
- virtual reality games arm (Experimental): Ten technological treatment sessions divided into 2 training sessions per week for 5 weeks.
  Interventions: Other: virtual reality games intervention
- robotic treadmill arm (Experimental): Ten traditional physical treatment sessions divided into 2 training sessions per week for 5 weeks.
  Interventions: Other: robotic treadmill intervention

INTERVENTIONS:
Other: traditional rehabilitation — Each session will include 50 minutes of traditional physical rehabilitation therapy
  Arms: control group
Other: virtual reality games intervention — Each session will include 30 minutes of traditional physical rehabilitation therapy followed by 20 minutes of robotic training by Tymo system (Tyromotion, Austria), a wireless platform for the balance and the postural control training that simulates floor walking and stairs climbing. Tymo system is connected to a screen and provides virtual reality games, adaptable to the functional capacity of the patient. Through the games proposed, the physiotherapist will decide to work in a dimension (antero-posterior or medio-lateral dimension) or in two dimensions (combining the antero-posterior and medio-lateral movements).
  Arms: virtual reality games arm
Other: robotic treadmill intervention — Each session will include 30 minutes of traditional physical rehabilitation therapy followed by 20 minutes of robotic training by Walker view (TecnoBody, Italy), a treadmill equipped with a sensorized belt with eight load cells and a 3D camera.to detect length, speed and symmetry of the pace and load, range of the trunk, hips and knees. Patients will be asked to walk at a comfortable speed, while the physiotherapist will be able to work on different parameters such as step length, load distribution, and step height. The setting will take place taking into account the clinical conditions of each patient, customizing the intervention. The Walker View will offer visual and auditory feedback to the patient, so as to correct gait in real time.
  Arms: robotic treadmill arm

SUMMARY:
The final goals of the present study is to propose a new approach in the hip fracture rehabilitation in elderly subjects, focused on the use of robotic device and to check the results not only at the end of the treatment but also in the long term, foreseeing 3 follow-up.

DETAILED DESCRIPTION:
Balance and deficit in walking are some of the main characteristics of aging and are considered among the risk factors for falls. Falls are a risk factor for future falls and are associated with other adverse health outcomes such as fear of falling or fractures. In particular, hip fracture in aged patients is an important health problem. In fact, one in three patients dies within the first year after injury, while survivors have poor quality of life For this reason, the development of prevention tools and innovative strategies in the rehabilitation field should be one of the main objectives in the treatment of the diseases afflicting the elderly, such as hip fractures. Effective interventions to promote hip recovery post hip fracture are characterized by intensive and repetitive movements. One treatment approach to increase number of steps during rehabilitation sessions and to improve the balance and the endurance of the patients is the use of robotic systems.

This study is a randomized controlled trial. A total of 195 patients with hip fractures will be recruited and randomly divided into three groups, to receive a traditional rehabilitation program or a robotic rehabilitation in addition to the traditional therapy. Assessments will be performed at baseline, at the end of treatment and 6 months, 1 year and 2 years from the end of the treatment. For the study, post-hospitalization subjects will be taken into consideration, after four weeks from the hospitalization. A 20 treatment sessions will be conducted, divided into 3 training sessions per week, for 7 weeks. The control group will perform traditional therapy sessions lasting 50 minutes. The technological intervention group will carry out 30 minutes of traditional therapy and 20 minutes of treatment with a robotic system.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to consent
* Traumatic event within 60 days
* Romberg test: negative
* Functional Ambulation Category (FAC) score ≤ 2
* Ranking scale score ≤ 3;

Exclusion Criteria:

* Past history of syncopal episodes
* Presence of non-pharmacologically compensated behavioral syndromes
* Presence of pain that prevents walking or standing
* Presence of neurological pathologies that compromise balance (Multiple sclerosis, Parkinson's disease, stroke, ataxias, poliomyelitis)
* Spinal stenosis
* Radiculopathy
* Neuropathies lower limbs
* Disabling disabilities that impair walking (eg congenital malformations of the foot)
* Heterometry > 2 cm
* Clinical dementia rating (CDR) score ≥ 3
* Severe systemic diseases with life expectancy < 1 year
* Patients unable to follow up.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
difference in falling risk among virtual reality games arm, robotic treadmill arm and control arm | before treatment, and 5 weeks, 6 months, 12 months and 24 months after intervention commencement
  falling risk will be evaluated by the Tinetti performance oriented mobility assessment (POMA). POMA test has two subscales, Balance and Gait sections. Total score is obtained by adding the scores of the two subscales (balance + gait) . Total score < 19 high fall risk, total score 19-24 medium fall risk, total score 25-28 low fall risk

SECONDARY OUTCOMES:
difference in gait performance among virtual reality games arm, robotic treadmill arm and control arm | before treatment, and 5 weeks, 6 months, 12 months and 24 months after intervention commencement
  gait performance will be evaluated by the walking speed evaluated by instrumental gait analysis
difference in fear of falling among virtual reality games arm, robotic treadmill arm and control arm | before treatment, and 5 weeks, 6 months, 12 months and 24 months after intervention commencement
  fear of falling will be evaluated by the Falls Efficacy Scale - International (FES-I). Higher scores represent greater the fear of falling (ranging from 16 to 64)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Riccardi, Principal Investigator — IRCCS-INRCA
Locations (2):
- Italy (2):
  - INRCA Research Hospital, Ancona
  - INRCA Research Hospital, Fermo

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134
- [Derived] Maranesi E, Riccardi GR, Lattanzio F, Di Rosa M, Luzi R, Casoni E, Rinaldi N, Baldoni R, Di Donna V, Bevilacqua R. Randomised controlled trial assessing the effect of a technology-assisted gait and balance training on mobility in older people after hip fracture: study protocol. BMJ Open. 2020 Jun 15;10(6):e035508. doi: 10.1136/bmjopen-2019-035508. PMID 32546491